CLINICAL TRIAL: NCT03718520
Title: The Influence of in Utero Cannabis Exposure on Neonatal Brain Morphology and Structural Connectivity
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-0004; R21DA043833 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Cannabis Use Disorder; PREG1; Drug Use; Fetal Exposure During Pregnancy; Neurodevelopmental Abnormality
Keywords: cannabis; fetal programming; pregnancy; infant neuroimaging
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal urine at 28-36 weeks gestation; maternal plasma and urine at delivery; neonate urine, meconium, cord blood and cord segment shortly after birth; maternal urine at 2 weeks postpartum; maternal urine at 1 year postpartum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prenatal exposed to cannabis: 50 mother-infant pairs with self-reported maternal chronic cannabis use during pregnancy
  Interventions: Other: no intervention, this is a purely observational study
- prenatal not-exposed to cannabis: 60 mother-infant pairs with no self-reported maternal cannabis use during pregnancy
  Interventions: Other: no intervention, this is a purely observational study

INTERVENTIONS:
Other: no intervention, this is a purely observational study — No intervention

SUMMARY:
Cannabis is the most commonly used drug by women during pregnancy with an estimated prevalence of use in Colorado of 5.7%. THC and its metabolites freely cross the placenta and blood-brain barrier to bind with cannabinoid receptors, disrupting the endogenous cannabinoid signaling system during a critical period of development of cortical circuitry structure and function. The density of cannabinoid receptors in the developing brain is high, especially in the limbic areas and prefrontal lobes. Research in animal models suggests synaptic plasticity in the prefrontal lobes as well the amygdala and hippocampus are impacted by the prenatal cannabis exposure; regions associated with both cognitive and emotional control, thus influencing long-term deficiencies in attention and impulsivity. This pilot study will collect preliminary data on the structural impact of in utero cannabis exposure on region-specific morphology and structural connectivity of white matter tracts that connect to the prefrontal lobes and the limbic regions shortly after birth, before confounding by the postnatal environment becomes a major influence.

DETAILED DESCRIPTION:
Cannabis is the most commonly used psychoactive substance among pregnant women, with an estimated prevalence of use between 5 to 20% in in the United States. Little is known about the neurodevelopmental consequences for the fetus, particularly in the context of contemporary cannabis use patterns including high potency strains, cannabinoids and novel routes of administration. Colorado leads the nation in implementation of legalized medical and retail marijuana. Coupled with a growing pro-marijuana advocacy movement, marijuana may be perceived as "safe" to use during pregnancy. The local actions of endocannabinoids are in place in the placenta during fetal brain development and THC and its metabolites freely pass the placental barrier and the fetal blood-brain barrier. Furthermore, cannabinoid receptors appear to be more widespread in the fetal and neonatal prefrontal cortex (PFC) and the limbic areas (the amygdala and hippocampus) than in the adult brain, thus the in utero period may be a sensitive period of human brain development during which exogenous cannabinoids could permanently alter neurodevelopmental processes. Human epidemiologic studies across diverse populations have reported an emerging theme of deficiencies related to impulse control and executive functioning among offspring with in utero exposure to cannabis starting in adolescence. Only rudimentary aspects of executive function are present in infants, thus evidence of an impact during infancy and the toddler years is sparse, inconsistent and confounded by the postnatal environment (i.e., daycare, caregiver functioning). Research is needed to evaluate the proximal impact of in utero cannabis exposure on robust metrics of neonatal brain morphology and structural integrity of white matter tracts that connect to the PFC and the limbic regions before the influence of postnatal exposures become a major confounding influence.

To address this challenge, a pilot prospective pre-birth cohort study will be conducted to investigate the impact of chronic in utero cannabis exposure by enrolling 110 mother-infant pairs (50 exposed and 60 unexposed controls) for a neonate neuroimaging scan within 2 weeks after birth. Chronic in utero cannabis exposure will be quantified using ultra-high performance liquid chromatography-tandem mass spectrometry (LC-MS) of neonatal meconium. The associations between in utero cannabis exposure and neural morphological outcomes will be examined by structural MRI and diffusion tensor imaging (DTI). The central hypothesis is that in utero cannabis exposure will be associated with alterations in grey and white matter development in the prefrontal lobe and its connectivity to limbic regions.

Specific Aim 1: To determine the magnitude of the association between in utero exposure to cannabis and neonate brain morphology and structural connectivity.

Hypothesis: In utero exposure to cannabis (assessed by THC metabolites in meconium) will be associated with the following neonate brain structural outcomes: (1) Grey matter: reduced volume in the PFC and limbic regions (i.e. the amygdala, hippocampus); (2) White matter: reduced structural integrity (assessed by fractional anisotropy) of white matter tracts that connect to the PFC and the limbic regions including the uncinate fasciculus and the cingulum bundle. The associations will be independent of other maternal substance use (i.e. tobacco), postnatal feeding practices (i.e. breastfeeding), socio-demographic characteristics and maternal mental health.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who are receiving prenatal care at the University of Colorado Hospital at Anschutz (UCH) or Denver Health Medical Center.
* maternal positive urine toxicology screen for cannabis at any clinical prenatal visit or self-report of cannabis during pregnancy at a clinical visit
* greater than ≥ 28 weeks gestation,
* aged ≥18 years,
* expecting a singleton birth,
* live in Colorado, and plan to deliver at UCH or Denver Health Medical Center .
* Inclusion criteria for unexposed controls will be identical to that of exposed cases with the exception that they cannot have a positive toxicology screen for cannabis or self-reported cannabis use during pregnancy.

Exclusion Criteria (for unexposed cases and controls):

* use of tobacco, alcohol or other drugs during pregnancy,
* serious chronic diseases (cancer, psychiatric diseases, steroid-dependent asthma, pre-existent diabetes mellitus of any kind),
* mothers who subsequently experience a fetal death or deliver a premature infant (< 37 weeks of gestation).
* Postnatal exclusions will include failure to collect meconium samples at birth, infant neurological trauma, other neurological conditions in the infant (e.g., epilepsy),
* suspicion of metal in body or other MRI contraindications in either the mother or infant.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — This study plans to enroll pregnant women.
Study Population: This will be an observational, pre-birth prospective pilot study of 110 mother-infant pairs (50 with prenatal cannabis exposure and 60 unexposed pairs) who deliver at two academic medical centers in the Denver Metro area of Colorado (Denver Health Medical Center and the University of Colorado Hospital at Anschutz. Unexposed controls will be frequency matched to exposed cases by maternal education level. To isolate the influence of cannabis exposure, mothers using tobacco, alcohol or other drugs during pregnancy will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
region specific grey matter volume (mm^2) in the PFC and limbic regions | 2 weeks postnatal age
  region specific volume (mm^2)
structural integrity measured by fractional anisotrophy of white matter tracks that connect the PFC and limbic regions | 2 weeks postnatal age
  mean fractional anisotrophy

SECONDARY OUTCOMES:
Negative affectivity based on a subscale from the Infant Behavioral Questionnaire (Rothbart, 1981) | 1 year postpartum
  Four subscales on the IBQ-R will be combined to form a negative affectivity scale including scales of Sadness, Distress to Limitations, Fear, and Falling Reactivity/Rate of Recovery from Distress.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Crume, PhD, MSPH, Principal Investigator — University of Colorado, Colorado School of Public Health
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No
A completely de-identified dataset will be created and may be shared upon PI-agreement ad development of data sharing agreements.